CLINICAL TRIAL: NCT04618289
Title: Effect of Vitamin D3-fortified Fruit Juice Supplementation on the Recovery of Iron Status in Childbearing-aged Women With Marginally Low Iron Stores
Brief Title: Effect of Vitamin D3-fortified Fruit Juice on Iron Status in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Dr Salma Faeza Ahmad Fuzi, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JKEUPM-2020-033
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Iron-deficiency
Keywords: iron status; hepcidin; vitamin D
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: A total of 120 participants who are eligible to continue with the study will be randomised to receive either 4000 IU (100 mcg) of vitamin D3-fortified fruit juice or placebo-fruit juice. The participants will be instructed to consume the vitamin D3-fortified fruit juice or placebo-fruit juice in the morning by diluting the powder in 150 ml of water, daily, for the 8-week duration of the study. All the participants will be reminded to not alter their dietary habits and physical activity, in addition, to abstaining from donating blood during the course of the study which may interfere with interpretation of study findings.
Who Masked: Participant, Investigator
Masking Description: The participants and researcher will be double-blinded as to which groups participants will be assigned. The researcher will administer the numbered supplement pot (i.e; 001) to the participants based on the sequence that participants attend their baseline clinic (Week 0). The blinding will be maintained throughout the study period of 8 weeks and allocation will not be unlocked until the end of the data analysis or during any adverse event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Group (Experimental): The vitamin D3-fortified fruit juice supplement that will be used is vitamin D3 cholecalciferol (4000 IU, 100 mcg, Fiatec Biosystem Sdn Bhd, Selangor, Malaysia).
  Interventions: Dietary Supplement: Vitamin D3-fortified fruit juice supplement
- Placebo Group (Placebo Comparator): The matching placebo will be also custom-produced and will be produced in the same manner, without the active ingredients by the same company. The placebo produced will match with vitamin D3 in terms of appearance, size, colour and taste to achieve the double-blind design.
  Interventions: Dietary Supplement: Vitamin D3-fortified fruit juice supplement

INTERVENTIONS:
Dietary Supplement: Vitamin D3-fortified fruit juice supplement — Vitamin D3-fortified fruit juice supplement

SUMMARY:
The present study is designed to utilise vitamin D3 supplements that may potentially act as an iron absorption enhancer to improve iron status in the Malaysian child-bearing aged women with low iron stores. In addition to investigating the efficacy, this study is also designed to assess the effect of a dose of vitamin D3 (4000 IU) on iron metabolism. The study will include the measurement of plasma hepcidin and 25(OH)D concentrations to investigate a possible mechanism that links vitamin D and iron deficiency, as postulated from the existing literature. For that reason, the aim of the study was to investigate the effect of an 8-week vitamin D3 supplementation on iron status indicators, including hepcidin concentration in childbearing aged Malaysian women with marginal iron stores. It is hypothesised that there will be a significant improvement in haematological indicators following 8-week daily vitamin D3 supplementation in the vitamin D group compared to placebo group. It is also hypothesised that plasma hepcidin concentration will be reduced following 8-week daily vitamin D3 supplementation, which results in increased iron stores.

DETAILED DESCRIPTION:
Anaemia is one of the most common micronutrient deficiencies worldwide and 50% of anaemia occurrences were reported to be caused by iron deficiency. The national prevalence of anaemia in Malaysia was 24.6%, which was higher in women (35.5%) compared to men (14.3%). Combatting anaemia/iron deficiency requires cohesive approach, as its occurrence is suggested to be multifactorial. Iron supplements have been widely used, whilst, either dietary pattern modification or iron fortification may be implemented at population levels. Despite numerous approach implemented, the problems are still prevalent. There is recently emerging evidence of the utilisation of vitamin D, as iron absorption enhancer that acts on suppression of hepcidin. However, there is scarcity of randomised controlled trial, investigating the effect of the vitamin D supplementation administered routinely, aiding as an iron absorption enhancer, on iron status especially in the general population, not only in Malaysia but worldwide.

This is a placebo controlled, double-blind randomised controlled trial, designed to investigate the effect of an 8-week vitamin D3-fortified fruit juice supplementation on haematological indicators and hepcidin response in a cohort of marginally-low iron stores Malaysia childbearing-aged women. The study is divided into 2 phases which includes Phase 1 when potential participants will be screened, randomised and Phase 2 where all the eligible participants will consume either vitamin D3-fortified fruit juices containing 4000 IU (100 mcg) (vitamin D) or placebo-fruit juices (placebo) daily for the duration of 8 weeks. At each 4-week interval, 10 ml fasted blood sample will be collected, as well as information on dietary habit and anthropometric measurement. Mixed model repeated measures analysis of variance (ANOVA) will be performed to determine the effect of intervention and the interaction with time points for all iron status and vitamin D status blood biomarkers. The clinical aspects of anticipated findings in the present study may be particularly applied to the recovery of iron status in iron deficient population, through the use of vitamin D supplementation in food fortification as a novel iron absorption enhancer.

ELIGIBILITY:
Inclusion Criteria:

* women of child bearing age
* healthy
* aged 19-40 years
* non-pregnant nor lactating.

Exclusion Criteria:

* had a history of gastrointestinal disorder (celiac disease, Crohn's disease, irritable bowel syndrome gastroesophageal reflux disease, peptic ulcers and other related gastrointestinal disorders which may cause nutrient malabsorption) and iron metabolic disorders such as iron overload
* had donated blood since the past 6 months
* regularly consuming nutritional supplements (iron, vitamin D, vitamin C, calcium).

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change of plasma ferritin concentration from baseline (week 0) to post intervention (week 8) | 3 time points (Week 0,4,8)
  Iron storage
Change of plasma hepcidin concentration from baseline (week 0) to post intervention (week 8) | 3 time points (Week 0,4,8)
  Iron regulator
Change of full blood counts concentration from baseline (week 0) to post intervention (week 8) | 3 time points (Week 0,4,8)
  Iron status

SECONDARY OUTCOMES:
Change of plasma 25(OH)D concentration from baseline (week 0) to post intervention (week 8) | 3 time points (Week 0,4,8)
  Circulating vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Salma Faeza Ahmad Fuzi, Principal Investigator — Dr
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmad Fuzi SF, Su Peng L, Zabaha Zalbahar N, Ab Manan N, Mohamad Alwi MN. Effect of vitamin D3-fortified fruit juice supplementation of 4000 IU daily on the recovery of iron status in childbearing-aged women with marginally low iron stores: Protocol for an 8-week, parallel group, double-blind randomized controlled trial. PLoS One. 2022 Mar 25;17(3):e0265772. doi: 10.1371/journal.pone.0265772. eCollection 2022. PMID 35333885